CLINICAL TRIAL: NCT04803890
Title: "No-Touch" Radiofrequency Ablation Using Octopus Electrodes and Combined RF Energy Delivery Mode for Small Hepatocellular Carcinoma (≤ 3cm): A Prospective Multicenter Study
Brief Title: "No-Touch" Radiofrequency Ablation for Small Hepatocellular Carcinoma (≤ 3cm): A Prospective Multicenter Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination d/t overlap with a new, extended protocol study.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2003-068-1108
Record Dates: First submitted 2020-03-31; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Radiofrequency Ablation; Microwave Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No touch radiofrequency ablation (Experimental): A total of 150 patients who have decided to participate in the study will be included, and prospective study will be performed to these patients for radio-frequency ablation using octopus electrodes, combined high-frequency transmission mode, and the 'No touch' technique.
  Interventions: Procedure: "No-Touch" Radiofrequency Ablation

INTERVENTIONS:
Procedure: "No-Touch" Radiofrequency Ablation — "No-Touch" Radiofrequency Ablation Using Octopus Electrodes and Combined RF Energy Delivery Mode

SUMMARY:
This study is a prospective multicenter study of the duration of treatment, the success rate, the frequency of complications, and the local recurrence rate of 12 months when Radio-frequency ablation therapy is performed for the treatment of HCC using the 'No touch' technique as a combined high-frequency transmission mode with Octopus electrodes. It aims to evaluate through. In addition, the results obtained from this prospective study were as follows: 1) Patients who underwent Radio-frequency ablation therapy by puncturing an existing tumor, and 2) Patients who underwent microwave ablation during the study period. The secondary goal is to evaluate which method is more effective in reducing the treatment time and recurrence rate compared to.

DETAILED DESCRIPTION:
1. Pre-treatment planning:

   The detailed plan of radio frequency ablation (RFA) will be implemented in accordance with the routine procedure of image evaluation prior to RFA. That is, after confirming the location of the tumor in the Multiphasic CT or MRI and evaluating the volume of the tumor and the relationship with adjacent blood vessels before RFA procedure, planning the insertion path and the number of ablation of the electrode for RFA, the recently used US- The CT-MR fusion tool is used to fuse the pre-treatment image and the ultrasound image to evaluate whether the tumor location on the ultrasound image matches the tumor found on the pre-treatment image. The location will be evaluated in real time. The end of the procedure is when an echo bubble of 5 mm to 10 mm or more is generated around the treated tumor, and it is confirmed that the enhancement of HCC disappears completely after RFA in immediate post procedure CT. In addition, if the boundary of the tumor is not well drawn on ultrasound, CEUS will be additionally used to confirm the location of the tumor. At this time, the ultrasonic fusion device to be used will be one of Phillips, GE, Samsung or Siemens' navigation systems available herein. The fused image guides the location of the electrodes to be installed in the tumor, the number of electrodes, and a safe access route.
2. RFA procedure As a device for RFA, a multi-viva generator and a separable clustered electrode (product name: Octopus electrode, Starmed Ltd), which are used herein, will be used.

   The procedure is to place the octopus high-frequency electrode in the periphery of the tumor (5 ± 2mm) using no touch technique under fusion ultrasound guidance, and then simultaneously apply high frequency to two electrodes up to 200W using the combined monopolar-bipolar mode with keeping the temperature at 90-100 degrees Celsius for about 5 to 30 minutes until the tumor and 5-10 mm echo band form around the tumor. During the RFA procedure, the US-CT-MR fusion tool (Navigator- GE & Siemens, Samsung) is used to fuse the pre-treatment image and the ultrasound image to match the echo bubble distribution and tumor location. It will be evaluated in real time.

   If the boundary of the tumor is unclear, it is difficult to grasp the boundary of the tumor 360 degrees as a whole, or if there is little normal tissue to install electrodes around the tumor, it is difficult to apply the No-touch technique. Therefore, in this study, the application rate of the No-touch technique will be evaluated among all recruited patients, and when evaluating the presence or absence of recurrence after the procedure, it is analyzed (intention to treat analysis) including puncture of the tumor, and treated with actual No-touch. It will be analyzed further.
3. Follow-up

   * CT (MRI if CT is contraindicated) will be performed immediately after RFA therapy as previously performed as a clinical routine, and it will be evaluated whether complete necrosis of the treated tumor has been achieved. If residual masses are identified or insufficient safety margins are not secured, additional procedures are performed and evaluated.
   * Alternatively, AFP or CEA, CBC, LFT and CT or MRI are performed 1 to 3 months after RFA procedure.
   * The follow up method is the same as the existing method, and blood tests and CT or MRI tests are performed every 3 to 4 months for 3 to 4 times during 12 months. This is due to the fact that most local recurrence occurs within 12 months, and the local recurrence rate will be evaluated based on this.
   * The final point of time for this study is based on the follow-up findings obtained at 12 ± 1 month after the procedure (short-term relapse rate evaluation).
   * However, after that, the patient will continue to perform CT or MR follow-up every 3 to 6 months until 2 years according to the routine follow-up protocol of the patient who has undergone existing RFA therapy.
4. Control group Of the patients who underwent RFA therapy for the treatment of HCC for a period of 2 years from 2018 to 2020, the patient group had been treated with conventional RFA and microwave ablation were enrolled. After performing the propensity score matching analysis using variables of age, gender, tumor size, tumor location, and liver function values, the same number of controls are selected and set.

ELIGIBILITY:
Inclusion Criteria:

* Agree to the protocol's requirements and submit a consent form
* 20 years old-85 years old
* Child-Pugh Class A or B7
* Among patients with cirrhosis, patients with hepatocellular carcinoma having a size of 1 cm-3 cm suspected of MDCT or MRI performed within 60 days are considered for radio-frequency ablation
* Patients who do not have a history of treatment for previous hepatocellular carcinoma, or who have a history of treatment for previous hepatocellular carcinoma, if recurrence has not been confirmed for at least 2 years after treatment

Exclusion Criteria:

* the number of liver tumors is 3 or more
* the maximum size of the tumor exceeds 3 cm
* diffuse infiltrative type
* the tumor adheres to the portal vein or hepatic vein or biliary tract of 5 mm or more
* patients with previous medical history of hepatocellular cancer who have recurrent hepatocellular cancer within 2 years
* the tumor is not visible even under CEUS-fusion image guidance
* Child-Pugh class B8 or C
* in case of invasion of liver vessels due to malignant hepatocellular carcinoma
* severe coagulopathy
* multiple distant metastasis
* the situation where the probability of obtaining appropriate data suitable for the research purpose is very low

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Local tumor progression (LTP) rate | 12 months after RFA
  No. of participants with LTP/ No. of participants receiving RFA

SECONDARY OUTCOMES:
Intrahepatic distant recurrence (IDR) rate | 12 months after RFA
  No. of participants with IDR/ No. of participants receiving RFA
Complication rate | 12 months after RFA
  No. of procedure-related complication/No. of participants receiving RFA

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No